CLINICAL TRIAL: NCT01911104
Title: Investigating the Underlying Mechanisms of Exercise Resistance in Individuals With Type 2 Diabetes
Brief Title: Exercise Resistance in Type 2 Diabetes
Acronym: RESIST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRIMDFH 471035; 471035 (Other: Florida Hospital IRB)
Record Dates: First submitted 2013-07-23; First posted 2013-07-30 (Estimated); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes
Keywords: muscle; mitochondrial function; exercise resistance; human; myotubes; epigenetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): 10 weeks of aerobic exercise
  Interventions: Behavioral: Exercise
- Active Control (No Intervention): Young athletes as a trained control

INTERVENTIONS:
Behavioral: Exercise — 10 weeks of aerobic exercise
  Arms: Exercise

SUMMARY:
The purpose of this study is to collect data to help researchers identify factors that prevent certain individuals from receiving the beneficial effects of exercise.

DETAILED DESCRIPTION:
STUDY OBJECTIVES/ENDPOINTS

1. The primary endpoint of the study is the maximal capacity for mitochondrial ATP synthesis measured using 31P magnetic resonance spectroscopy (MRS).
2. The principal secondary endpoint is the relationship between exercise-induced changes in mitochondrial function in vivo and exercise mimetic-induced changes in mitochondrial function in vitro.
3. The principal tertiary endpoint is the relationship between the basal promoter methylation status of key genes involved in fuel metabolism and known to be activated by exercise in skeletal muscle tissue and cells and the exercise-induced response in mitochondrial function.

As exercise has an array of metabolic effects, and we are well positioned with our cutting-edge methodologies here at the Translational Research Institute (TRI), we will also measure whole body insulin sensitivity and metabolic flexibility by hyperinsulinemic-euglycemic clamp, substrate oxidation and energy expenditure in the whole room calorimeter/metabolic chamber and intramyocellular lipid content.

ELIGIBILITY:
Type 2 Diabetes Inclusion Criteria (Group 1)

* Age 30 to 65 years.
* Male and Female
* Type 2 diabetes determined by self-report or by a fasting glucose > 126mg/dl
* POCT HbA1c result is 5.7-8.8% or for those on anti-diabetic medications, POCT HbA1c < 8.9% (no lower limit defined to account for those who illustrate tight glycemic control due to anti-diabetic medications).
* HbA1c between 6.0% and 8.5% or for those on anti-diabetic medications, HbA1c ≤ 8.5% (no lower limit defined to account for those who illustrate tight glycemic control due to anti-diabetic medications). If a participant misses the screening HbA1c by a small margin (HbA1c ± 0.1%), the HbA1c can be repeated once.
* Not involved in regular exercise program
* Willing to exercise every day for the study period
* If applicable, those currently taking anti-diabetic medication are taking metformin, a sulfonylurea, DPP IV inhibitor, alpha-glucosidase inhibitor, a meglitinide, colesevelam, cycloset or a SGLT2 inhibitor. Those taking 2 of these medications may proceed.
* If applicable, willing to cease anti-diabetic medication use for the duration of the intervention.
* BMI ≥ 22 kg/m2

Young Athletes Inclusion Criteria (Group 2)

* Age 18 to 50 years
* Male and Female
* Engaged in a minimum of 4 cumulative hours of moderate to vigorous intensity aerobic exercise, over a minimum of 3 days per week.
* BMI between 18 and 29.9 kg/m2
* VO2max > 45 ml/min/kg BW

Non-diabetes Inclusion Criteria (Group 3)

* Age 30 to 65 years
* Male and Female
* Not involved in a regular exercise program
* Willing to exercise every day for the study period
* BMI ≥ 22 kg/m2

General Exclusion Criteria A=all groups, Ex=exercise group only, ND=Non-diabetes group only

* Resting blood pressure ≥ 160/100 mm Hg (A)
* Triglycerides > 500 mg/dL (A)
* HbA1c ≥ 6.5% (ND)
* Previous or current use of an insulin pump or multiple insulin injections per day or any diabetes medications that the participant cannot refrain from for the duration of the study. (A)
* Treatment with thiazolidinediones (TZDs) or GLP-1 agonists within the last 3 months. (A)
* Unable or unwilling to communicate with staff or to provide written informed consent. (A)
* Failure to complete baseline testing. (A)
* Not physically capable of performing the exercise required of the study protocols. (Ex)
* Consuming >14 alcoholic beverages per week. (A)
* Plans to be away >2 weeks in the next 3 months. (A)
* Lack of support from primary health care provider and/or family members.(Ex)
* Significant weight loss in the past year (>20 lbs) or current use of weight loss medications. (A)
* Bariatric surgery or planning bariatric surgery in the next 6 months.(Ex)
* Presence of clinically significant abnormalities on ECG (A)
* Any renal, cardiac, liver, lung, or neurological disease that in the opinion of the Investigator would compromise participant safety (A)
* Use of drugs known to affect energy metabolism or body weight: including, but not limited to: orlistat, sibutramine, ephedrine, phenylpropanolamine, corticosterone, etc (A)
* Current treatment with blood thinners or anti-platelet medications that cannot be safely stopped for testing procedures. (A)
* New onset (<3 months on a stable regime) hormone replacement therapy. (A)
* Current use of beta-adrenergic blocking agents (A)
* Alcohol or other drug abuse (A)
* Current smokers (smoking within the past 3 months) (A)
* Gait problems (Ex)
* Unwilling or unable to abstain from caffeine, alcohol or strenuous exercise (48h) prior to metabolic rate measurements (A)
* Increased liver function tests (AST/ALT/GGT/or alkaline phosphatase greater than 2.5 times the upper limit of normal) (A)
* Metal objects that would interfere with the measurement of body composition /MRS such as implanted rods, surgical clips, etc (A)
* Any NYHA class of CHF (A)
* Abnormal blood count/Anemia, blood transfusion or blood donation within the last 2 months. (A)
* Major surgery on the abdomen, pelvis, or lower extremities within previous 3 months (A)
* Bariatric surgery or liposuction within the previous 3 years (Ex)
* Cancer (active malignancy with or without concurrent chemotherapy) (A)
* Rheumatoid disease (A)
* Bypass graft in limb (A)
* Known genetic factor (Factor V Leiden, etc) or hypercoagulable state (A)
* Peripheral neuropathy, involving more than the toes (A)
* Claustrophobia (A)
* Major Depression (Ex)
* Presence of an eating disorder or eating attitudes/behaviors that could interfere with the study completion (Ex)
* Females that are currently or have been pregnant or are currently or have nursed a child within the last 12 months (A)
* Presence of any condition that, in the opinion of the investigator, compromises participant safety or data integrity or the participants' ability to complete the training protocol (Ex).

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-10-31 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in ATPmax | Baseline and 10 weeks
  The primary endpoint of the study is the maximal capacity for mitochondrial ATP synthesis (ATPmax) measured using 31P magnetic resonance spectroscopy (MRS).

SECONDARY OUTCOMES:
Change in in vivo and in vitro mitochondrial function | Baseline and 10 weeks
  The principal secondary endpoint is the relationship between exercise-induced changes in mitochondrial function (ATPmax) in vivo and exercise mimetic-induced changes in mitochondrial function in vitro (maximal oxygen consumption of the human primary myotubes by the Oroboros® oxygraph).

OTHER OUTCOMES:
Promoter methylation | Baseline
  The principal tertiary endpoint is the relationship between the basal promoter methylation status of key genes involved in fuel metabolism and known to be activated by exercise in skeletal muscle tissue and cells and the exercise-induced response in ATPmax.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M Sparks, PhD, Principal Investigator — Translational Research Institute for Metabolism and Diabetes
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

REFERENCES:
- [Derived] Whytock KL, Pino MF, Sun Y, Yu G, De Carvalho FG, Yeo RX, Vega RB, Parmar G, Divoux A, Kapoor N, Yi F, Cornnell H, Patten DA, Harper ME, Gardell SJ, Smith SR, Walsh MJ, Sparks LM. Comprehensive interrogation of human skeletal muscle reveals a dissociation between insulin resistance and mitochondrial capacity. Am J Physiol Endocrinol Metab. 2023 Oct 1;325(4):E291-E302. doi: 10.1152/ajpendo.00143.2023. Epub 2023 Aug 16. PMID 37584609
- [Derived] Carnero EA, Bock CP, Distefano G, Corbin KD, Stephens NA, Pratley RE, Smith SR, Goodpaster BH, Sparks LM. Twenty-four hour assessments of substrate oxidation reveal differences in metabolic flexibility in type 2 diabetes that are improved with aerobic training. Diabetologia. 2021 Oct;64(10):2322-2333. doi: 10.1007/s00125-021-05535-y. Epub 2021 Aug 17. PMID 34402932
- [Derived] Pino MF, Stephens NA, Eroshkin AM, Yi F, Hodges A, Cornnell HH, Pratley RE, Smith SR, Wang M, Han X, Coen PM, Goodpaster BH, Sparks LM. Endurance training remodels skeletal muscle phospholipid composition and increases intrinsic mitochondrial respiration in men with Type 2 diabetes. Physiol Genomics. 2019 Nov 1;51(11):586-595. doi: 10.1152/physiolgenomics.00014.2019. Epub 2019 Oct 7. PMID 31588872